CLINICAL TRIAL: NCT03080662
Title: Impact of Inspiratory Muscle Training on Daily Physical Activity (INAF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Diego Agustín Rodríguez, Principal Investigator, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INAF
Record Dates: First submitted 2017-03-07; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Inspiratory Muscle Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham valve (Placebo) (Sham Comparator): Sham Inspiratory valve (without resistance)
  Interventions: Device: ORYGEN DUAL Sham Valve
- Intervention (Experimental): Inspiratory valve with increase resistance
  Interventions: Device: ORYGEN DUAL Valve

INTERVENTIONS:
Device: ORYGEN DUAL Sham Valve — Training of the inspiratory muscles during 5 weeks
  Arms: Sham valve (Placebo)
Device: ORYGEN DUAL Valve — Training of the inspiratory muscles during 5 weeks
  Arms: Intervention

SUMMARY:
The impact of the reduction of daily physical activity (DPA) in patients with COPD (chronic obstructive pulmonary disease) is a highly studied area, due to its impact on the quality of life and the clinical evolution of the disease . This fact has multifactorial components: its function is naturally diminished with time, and its effects on the loss of physical condition (decondition). However, dynamic hyperinflation and respiratory muscular dysfunction, especially in patients with more symptomatology, have been identified as those that have the most relevant factors that impact on daily physical activity Due to the detrimental effects of the pulmonary hyperinflation, the diaphragm is flatter and shorter, being in a position of mechanical disadvantage. This contributes to a reduced effort capacity and increase in the dyspnea of patients during daily activities.

Resistance training improves their exercise capacity and reduces dyspnea, however it does not improve inspiratory muscle strength. It is for this reason, that specific training of the inspiratory muscles, offers special interest in patients with decreased inspiratory muscle strength and pulmonary hyperinflation.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the respiratory rehabilitation programme participants must have stable COPD (at least 4 weeks), inspiratory muscle weakness (PImax <70%) and pulmonary hyperinflation (TLC > 120%). Patient that have signed inform consent.

Exclusion Criteria:

* Hospitalization within the previous 14 days
* Current participation in rehabilitation program,
* Locomotor or neurological condition or disability limiting the ability to perform exercise,
* Lung transplantation or lung volume reduction surgery foreseen within 1 month after discharge.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01-22 (Actual); Primary Completion 2017-12-15 (Estimated); Study Completion 2018-03-15 (Estimated)

PRIMARY OUTCOMES:
improvement of daily physical activity | Baseline and 5 weeks
  Change From Baseline at least 10% moderate to vigorous daily physical activity measured by accelerometer

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Del Mar, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No